CLINICAL TRIAL: NCT01226095
Title: A Prospective, Multi-center, Post-marketing Observational Study to Evaluate the Effectiveness and Compliance of Ibuprofen in a Sustained Release Form in the Treatment of Egyptian Osteoarthritic Patients
Brief Title: Evaluation of the Effectiveness, Compliance of Ibuprofen in a Sustained Release Form in the Treatment of Egyptian Osteoarthritic Patients
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Clintek (Unknown)
Responsible Party: Sponsor
Other Study IDs: P12-162
Record Dates: First submitted 2010-09-07; First posted 2010-10-21 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2012-01

CONDITIONS: Osteoarthritis; Pain; Morning Stiffness
Keywords: Osteoarthritis; Pain; Morning stiffness
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Osteoarthritic patients: Patients male or female, age ≥ 18 having clinical or radiological evidence of osteoarthritis

SUMMARY:
This is a prospective, multi-center, post-marketing observational study to evaluate the effectiveness and compliance of ibuprofen in a sustained release form in the treatment of Egyptian osteoarthritic patients.

DETAILED DESCRIPTION:
This was a prospective, longitudinal, multicenter observational study conducted in a clinical practice setting where the study product was used in osteoarthritis patients as indicated in the approved package insert; the dosing regimen of Brufen retard is 2 tablets as a single dose once daily.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking treatment for osteoarthritis and there are clinical or radiological evidence of the disease,
* Male or female, age ≥ 18
* Designated to treatment with Ibuprofen in a sustained release form (Brufen Retard) according to the best criterion of the physician and if he decides to treat the patient according to labeled indication and dose for 4 weeks.
* Patients who have given their written informed consent to participate in the study
* Patients who are currently taking non steroidal anti inflammatory drugs (NSAIDs), should complete an initial washout phase 10 days depending on the half life of the drug taken

Exclusion Criteria:

* Contraindications as described in company core data sheet (CCDS) and specifically
* Patients with active peptic ulcer
* Patients who have presented reactions of hypersensitivity (asthma , rhinitis or urticaria ) with ibuprofen or other anti-inflammatory non steroids
* Patients with active cardiovascular disease and those taking aspirin/warfarin for prophylaxis for myocardial infarction (MI) or stroke
* Patients with moderate to severe renal diseases
* Patients with moderate to severe hepatic disease
* Patients with Crohn's disease
* Patients included currently in another study
* Women of childbearing potential must not be pregnant
* Any patients the investigators consider ineligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Eldessouky, MBBC, Study Director — Abbott (Egypt)
Locations (15):
- Egypt (15):
  - Site Reference ID/Investigator# 42584, Alexandria
  - Site Reference ID/Investigator# 42585, Alexandria
  - Site Reference ID/Investigator# 42591, Alexandria
  - Site Reference ID/Investigator# 42593, Alexandria
  - Site Reference ID/Investigator# 42594, Alexandria
  - Site Reference ID/Investigator# 29755, Cairo
  - Site Reference ID/Investigator# 42582, Cairo
  - Site Reference ID/Investigator# 42583, Cairo
  - Site Reference ID/Investigator# 42586, Cairo
  - Site Reference ID/Investigator# 42587, Cairo
  - Site Reference ID/Investigator# 42588, Cairo
  - Site Reference ID/Investigator# 42589, Cairo
  - Site Reference ID/Investigator# 42590, Cairo
  - Site Reference ID/Investigator# 42592, Cairo
  - Site Reference ID/Investigator# 42595, Cairo

RESULTS

PARTICIPANT FLOW:
Groups:
- Brufen Retard: Male or female participants ≥ 18 years of age in Egypt with osteoarthritis who took Brufen Retard (open-label ibuprofen in a sustained release form) administered per the Prescribing Information for 4 weeks.
Period: Overall Study
Arm/Group | Brufen Retard
Started | 519
Completed | 518
Not Completed | 1
Not completed — Poor compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brufen Retard
Number analyzed (Participants) | 519
Age Continuous [Mean (Standard Deviation); unit: years] | 54.66 (10.36)
Age Continuous [Median (Full Range); unit: years] | 55 [23 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 348
  Male | 171
Region of Enrollment [Number; unit: participants]
  Egypt | 519

OUTCOME MEASURES:

1. Primary Outcome: Day and Night Mean Pain Score for the Previous 24 Hours on a Nine-point Scale (0 = no Pain to 8 = Very Severe Pain) at Visit 3 (4 Weeks Following Treatment) in Comparison to Baseline.
Description: Scoring of day and night pain for the previous 24 hours was performed on a nine-point scale (0 = no pain to 8 = very severe pain) at each visit and compared to baseline. The overall mean pain score was calculated for participants who completed the study at each visit.
Time Frame: Baseline and 4 weeks
Population: Effectiveness data were analyzed using the intent-to-treat (ITT) and per-protocol (PP) populations, each of which consisted of all 519 enrolled participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Brufen Retard Baseline (Visit 1): Male or female participants ≥ 18 years of age in Egypt with osteoarthritis prior to administration of Brufen Retard (open-label ibuprofen sustained release form) at Baseline per the Prescribing Information.
- Brufen Retard (Visit 3, Week 4): Male or female participants ≥ 18 years of age in Egypt with osteoarthritis who took Brufen Retard (open-label ibuprofen in a sustained release form) administered per the Prescribing Information for 4 weeks.
Arm/Group | Brufen Retard Baseline (Visit 1) | Brufen Retard (Visit 3, Week 4)
Number analyzed (Participants) | 519 | 519
units on a scale | 6.12 (1.38) | 2.10 (1.70)
Statistical Analysis 1: Comparison: Brufen Retard Baseline (Visit 1) vs Brufen Retard (Visit 3, Week 4); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Percent of Participant Compliance
Description: The frequency with which the participant forgot to take treatment or changed dose/administration was determined by comparing the actual number of tablets taken by the participant to the scheduled number of tablets since the last visit. Results are presented in percent (0 - 100% scale, with 100% being perfect compliance and 0% being no compliance at all).
Time Frame: 2 and 4 weeks
Population: Compliance was calculated for all participants using the dose actually taken and the dose that should have been taken.
Measure: Number; unit: percentage of participant compliance
Groups:
- Brufen Retard (Visit 2, Week 2): Male or female participants ≥ 18 years of age in Egypt with osteoarthritis who took Brufen Retard (open-label ibuprofen in a sustained release form) administered per the Prescribing Information for 2 weeks.
- Brufen Retard (All Visits): Male or female participants ≥ 18 years of age in Egypt with osteoarthritis who took Brufen Retard (open-label ibuprofen in a sustained release form) administered per the Prescribing Information throughout this post-marketing observational study.
Arm/Group | Brufen Retard (Visit 2, Week 2) | Brufen Retard (Visit 3, Week 4) | Brufen Retard (All Visits)
Number analyzed (Participants) | 519 | 519 | 519
percentage of participant compliance | 99.39 (0.99) | 97.71 (2.41) | 98.55 (1.86)

3. Secondary Outcome: Number of Participants With Joint Tenderness/Stiffness at Each Visit
Description: Joint tenderness/stiffness was measured using a 4-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) at each visit.
Time Frame: Baseline, 2 weeks, and 4 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Brufen Retard Baseline (Visit 1) | Brufen Retard (Visit 2, Week 2) | Brufen Retard (Visit 3, Week 4)
Number analyzed (Participants) | 519 | 519 | 519
participants
  No joint tenderness/stiffness | 17 | 87 | 262
  Mild joint tenderness/stiffness | 75 | 271 | 210
  Moderate joint tenderness/stiffness | 261 | 156 | 44
  Severe joint tenderness/stiffness | 166 | 5 | 3

4. Secondary Outcome: Number of Participants Who Improved (Reduced), Had no Change (Equal at Baseline and Visit), and Worsened (Increased) in Joint Tenderness/Stiffness at Visit 2 (After 2 Weeks of Treatment) and Visit 3 (After 4 Weeks of Treatment).
Description: Duration of morning stiffness at each visit was assessed and the number of participants who improved, had no change, or worsened at each visit, following 2 and 4 weeks of treatment (Visit 2 and Visit 3, respectively) was calculated.
Time Frame: 2 and 4 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Brufen Retard (Visit 2, Week 2) | Brufen Retard (Visit 3, Week 4)
Number analyzed (Participants) | 519 | 519
Participants
  Improved | 410 | 473
  No change | 109 | 46
  Worsened | 0 | 0

5. Secondary Outcome: Duration of Morning Stiffness
Description: The duration of morning stiffness in minutes was assessed at each visit.
Time Frame: Baseline, 2 weeks, and 4 weeks
Population: Effectiveness data were analyzed using the intent-to-treat (ITT) and per-protocol (PP) populations, however, only participants with available morning stiffness data were included in the analysis for each visit.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Brufen Retard Baseline (Visit 1) | Brufen Retard (Visit 2, Week 2) | Brufen Retard (Visit 3, Week 4)
Number analyzed (Participants) | 493 | 487 | 480
minutes | 24.20 (15.68) | 13.49 (11.67) | 7.76 (9.56)

6. Primary Outcome: Number of Participants Who Improved (Reduced Pain), Had no Change (Equal Scores at Baseline and Visit), and Worsened (Increased Pain) at Visit 3 (After 4 Weeks of Treatment).
Description: Scoring of day and night pain for the previous 24 hours was performed on a 9-point scale (0 = no pain to 8 = very severe pain) at each visit. The number of participants at Visit 3 (after 4 weeks of treatment) who improved (had reduced pain; from higher baseline score to lower Visit 3 score), had no change (equal scores at baseline and Visit 3), and worsened (increased pain; from lower baseline score to higher Visit 3 score) was calculated.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Brufen Retard (Visit 3, Week 4)
Number analyzed (Participants) | 519
Participants
  Improved | 516
  No change | 3
  Worsened | 0

7. Secondary Outcome: Number of Participants With 80% Reduction From Baseline in Duration of Morning Stiffness at Visit 2 (2 Weeks of Treatment) and Visit 3 (4 Weeks of Treatment)
Description: The number of participants who achieved an 80% reduction from baseline in morning stiffness was calculated at each visit.
Time Frame: 2 and 4 weeks
Population: Data were analyzed for all participants for which data were available.
Measure: Number; unit: participants
Arm/Group | Brufen Retard (Visit 2, Week 2) | Brufen Retard (Visit 3, Week 4)
Number analyzed (Participants) | 487 | 480
participants
  Achieved 80% reduction in morning stiffness | 58 | 211
  Did not achieve 80% reduction morning stiffness | 429 | 269

8. Secondary Outcome: Number of Participants With the Ability to Carry Out Normal Activities at Each Visit
Description: The number of participants who were able or unable to carry out normal activities was assessed at each visit.
Time Frame: Baseline, 2 weeks, and 4 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Brufen Retard Baseline (Visit 1) | Brufen Retard (Visit 2, Week 2) | Brufen Retard (Visit 3, Week 4)
Number analyzed (Participants) | 519 | 519 | 519
participants
  Yes | 172 | 381 | 471
  No | 347 | 138 | 48

9. Secondary Outcome: Number of Participants Who Experienced Adverse Events and Serious Adverse Events
Description: Tolerability was assessed by collecting adverse events during the course of the study up to 30 days following the last dose of Brufen Retard. The number of participants experiencing a serious or non-serious adverse event is summarized. See the Reported Adverse Event section for details.
Time Frame: Baseline to 4 weeks
Population: The tolerability population included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Brufen Retard
Number analyzed (Participants) | 519
participants
  Serious adverse events | 0
  Non-serious adverse events | 41

ADVERSE EVENTS:
Time Frame: All adverse events that occurred during the course of the study were reported. Adverse events occurring during the study were reported up to 30 days after the last dose of open-label ibuprofen sustained release form.
Arm/Group | Brufen Retard
Serious Adverse Events (participants affected / at risk) | 0/519
Other Adverse Events (participants affected / at risk) | 41/519
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brufen Retard (N=519)
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 6
Gastritis (Gastrointestinal disorders) | 20
Gastrointestinal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Reflux oesophagitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 1
Headache (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection